CLINICAL TRIAL: NCT00671619
Title: A Phase I, Randomized, Vehicle-Controlled, Double-Blind, Mono-Centric, Single and Repeated Dose, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ESBA105 Eye Drops in Healthy Subjects
Brief Title: Study of ESBA105 Eye Drops in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ESBATech AG (Industry)
Responsible Party: Peter Lichtlen, Medical Director, ESBATech AG
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ESBA105CRD01
Record Dates: First submitted 2008-04-28; First posted 2008-05-05 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: opthalmology; antibody fragment; TNF alpha
MeSH Terms: interventions — ESBA105

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ESBA105 — eye drops

SUMMARY:
Objectives:

To evaluate the safety, tolerability and pharmacokinetics of ESBA105 administered topically to the eye for up to 28 days in healthy volunteers.

To determine the systemic exposure to ESBA105 upon single and repeated-dose topical application to the eye in healthy volunteers.

DETAILED DESCRIPTION:
ESBA105 is an anti TNF single chain antibody fragment

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian subjects.
* Written informed consent prior to any study procedures including screening tests for eligibility.
* Subjects should be in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Normal sitting blood pressure and pulse rate, i.e.: BP: 100-160 mm Hg systolic, 50-90 mm Hg diastolic and pulse rate: 45-100 bpm. Blood pressure and pulse will be measured after 3 minutes resting in a sitting position.
* Bilateral corrected visual acuity of at least 0.9
* No need for regular concomitant medication.
* Ability to communicate well with the investigator and comply with the requirements of the entire study.
* Use of qualified contraception

Exclusion Criteria:

* Any evidence of infectious disease as evidenced by medical history, clinical examination, positive serology results which indicate the presence of hepatitis B and/ or C or HIV infection or positive results of the QuantiFERON TB Gold test based latent tuberculosis testing.
* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of any allergy including allergic conjunctivitis requiring acute or chronic treatment (seasonal allergic rhinitis not associated to conjunctivitis which requires no treatment may be tolerated).
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Existence of any surgical or medical condition which might interfere with the evaluation of the general drug safety and tolerability including clinically relevant ophthalmological diseases, impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, haematological abnormalities, psychiatric diseases, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract.
* Shallow anterior chamber, closed angle glaucoma or any other contraindication to eye dilation for ophthalmological examination.
* History or presence of any other clinically relevant (in the opinion of the Investigator) ocular disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | several timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Pharma Contract, Basel, Switzerland